CLINICAL TRIAL: NCT04942509
Title: Coloring as a Brief Mindfulness-based Intervention for Stress Reduction Among Nurses
Brief Title: Mindful Coloring to Reduce Nurses' Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Janet Fong, Research Assistant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBRE-20-162
Record Dates: First submitted 2021-06-06; First posted 2021-06-28 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Stress (Psychology); Burn Out (Psychology)
Keywords: nurses; coloring; brief mindfulness-based intervention; mental well-being; mindfulness
MeSH Terms: conditions — Burnout, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants were allocated into the experimental and wait-list control groups. The experimental group colored for at least 5 days during a 10-day period while the control group did not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coloring (Experimental): This group did mindful coloring for at least 5 days or at least 100 minutes in total during a 10-day period
  Interventions: Behavioral: Coloring as a brief mindfulness-based intervention
- Wait-list control (No Intervention): This group did not do mindful coloring at all during a 10-day period.

INTERVENTIONS:
Behavioral: Coloring as a brief mindfulness-based intervention — Participants watched an instructional video on mindful coloring at the beginning of the intervention and colored mindfully for at least 5 days or 100 minutes in total during a 10-day period. The intervention included a coloring booklet that contained mandala patterns for coloring.
  Arms: Coloring

SUMMARY:
The purpose of this study was to investigate whether nurses who did mindful coloring for at least five working days during a 10-day period experienced stress reduction afterwards.

DETAILED DESCRIPTION:
Enrolled participants who met inclusion criteria (full-time clinical nurses working for at least five days during a specified 10-day period) were randomized in 1:1 ratio to the coloring or control groups. A third party did the allocation sequence and concealment. After giving informed consent, participants completed the baseline questionnaire and the coloring group watched an instructional video on mindful coloring. The coloring group were asked to color for any length of time on at least five working days during a 10-day period (period A) while the control group were asked to do it on a subsequent 10-day (period B). The post-intervention questionnaire was completed by both groups at the end of period A. The study was completed after period B.

ELIGIBILITY:
Inclusion Criteria:

* Full time clinical nurses working under the Hospital Authority who would be working for at least 5 days during a specified 10-day study period.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress | Time point 1: pre-intervention. Time point 2: post-intervention (10 days)
  Scores of 0-40 measured by the Perceived Stress Scale. A positive outcome is indicated by a lower post-intervention score.

SECONDARY OUTCOMES:
Change in mental well-being | Time point 1: pre-intervention. Time point 2: post-intervention (10 days)
  Scores of 7-35 measured by the short Warwick-Edinburgh Mental Well-being Scale. A positive outcome is indicated by a higher post-intervention score.
Change in burnout | Time point 1: pre-intervention. Time point 2: post-intervention (10 days)
  Three subscales (each with a separate score) assessing three facets of burnout including Emotional Exhaustion (scores 0-54), Depersonalisation (scores 0-30) and Personal Accomplishment (scores 0-48) measured by the Maslach Burnout Inventory - Human Services Survey for medical personnel. Burnout is represented by a combination of high emotional exhaustion and depersonalization scores, together with a low personal accomplishment score. Positive outcomes are indicated by a lower score in Emotional Exhaustion and Depersonalisation, and a higher score in Personal Accomplishment.
Change in trait mindfulness | Time point 1: pre-intervention. Time point 2: post-intervention (10 days)
  Scores of 24-120 measured by the Five Facets Mindfulness Questionnaire - short form. A positive outcome is indicated by a higher post-intervention score.

CONTACTS AND LOCATIONS:
Overall Officials: Shuk Yan Janet Fong, MSocSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Participants were ensured confidentiality in this study.

REFERENCES:
- [Derived] Fong JSY, Hui ANN, Ho KM, Chan AKM, Lee A. Brief mindful coloring for stress reduction in nurses working in a Hong Kong hospital during COVID-19 pandemic: A randomized controlled trial. Medicine (Baltimore). 2022 Oct 28;101(43):e31253. doi: 10.1097/MD.0000000000031253. PMID 36316873